CLINICAL TRIAL: NCT06418490
Title: Navigating the Biliary Maze：a Retrospective Cohort Study of Augmented Reality Improving Outcomes in Choledochal Dilation Resection
Brief Title: The Application of Digital Intelligent Diagnostic and Therapeutic Technology in Biliary Dilation Diagnosis
Acronym: DIIBD
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-042
Record Dates: First submitted 2024-04-24; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Congenital Biliary Dilatation; Choledochal Cyst
Keywords: Congenital Biliary Dilatation; Choledochal Cyst; Augmented reality; Digital intelligent; Three-dimensional visualization
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D-group: After adequate general anesthesia, the non-3D group underwent conventional choledochal cyst excision surgery, while the 3D group underwent choledochal cyst excision surgery guided by three-dimensional visualization technology or enhanced reality navigation.
  Interventions: Device: Three-dimensional visualization technology
- Non-3D Group: After adequate general anesthesia, the non-3D group underwent conventional choledochal cyst excision surgery, while the 3D group underwent choledochal cyst excision surgery guided by three-dimensional visualization technology or enhanced reality navigation.

INTERVENTIONS:
Device: Three-dimensional visualization technology — Three-dimensional reconstruction technology is a software that can collect CT and MRI data, perform image segmentation and three-dimensional reconstruction of the liver, gallbladder, dilated bile ducts, pancreas, venous, and arterial systems step by step. The software is called Abdominal Medical Image 3D Visualization Software (MI-3DVS, software copyright registration number: 2008SR18798).The AR-ANS (Software Copyright No.: 2018SR840555) is an intraoperative navigation system that integrates three-dimensional visualization technology.This modification provides visual guidance for surgeons when ligating or protecting critical vascular tissues during surgery.
  Other Names: Augmented Reality Navigation
  Groups: 3D-group

SUMMARY:
This research discusses the clinical application value of augmented reality navigation technology combined with three-dimensional visualization technology in improving surgical safety and promoting the development of precision surgery. This technology can reduce intraoperative vascular and bile duct injuries, effectively avoid serious postoperative complications, and reduce residual cysts.

DETAILED DESCRIPTION:
Choledochal cysts (CC) have traditionally been considered as cystic dilatations of the extrahepatic bile duct. Choledochal cysts are now referred to as choledochal dilatation, which also includes intrahepatic and extrahepatic cysts. Choledochal cysts are defined as cystic dilatations involving the bile duct tree of single or multiple segments of the intrahepatic and extrahepatic bile ducts. In 1959, Alonso-Lej et al. first divided CC into 3 types based on the location of bile duct dilatation. It was not until 1977 that Todani et al. revised the classification, adding 2 more types of CCs, which is the most commonly used classification by clinicians today; however, some experts dispute this, claiming that each type of CC has its own natural history, complications, and treatments. It is suggested to focus more on the pathogenesis rather than a simple anatomical classification of the bile duct tree. Choledochal cysts are a rare anomaly and are sometimes considered as a precancerous condition, which often leads to diagnostic challenges. The typical presentation of this condition is nonspecific. Medical teams must have a high clinical suspicion of choledochal cysts when investigating patients with jaundice, abdominal pain, and palpable abdominal masses. Due to the ambiguity of these symptoms and physical examination findings, appropriate imaging studies are crucial for diagnosis. Resection of choledochal dilatation has shown excellent results, with a complication-free rate of 89% and an overall 5-year survival rate exceeding 90%. Therefore, early diagnosis and appropriate management are essential to achieve optimal outcomes and a good prognosis.

Clinical practice has confirmed that the modern digital imaging technology, such as three-dimensional visualization and augmented reality navigation technology, built for hepatobiliary surgery diagnosis and treatment platform plays a crucial guiding role in precise preoperative assessment, lesion localization, formulation of optimal surgical plans, and intraoperative navigation to avoid collateral damage. Professor Fang Chihua's team has conducted long-term research and breakthroughs in this field. A significant portion of the literature in the field of digital intelligent diagnosis and treatment technology retrieved from SinoMed - China Biomedical Literature Service System comes from Professor Fang Chihua's team. The team has published consecutive expert consensus in the Chinese Journal of Practical Surgery in the field of digital intelligence in hepatobiliary surgery, including the publication of "Expert Consensus on Precise Diagnosis and Treatment of Three-Dimensional Visualization of Hepatobiliary Stones (2019 Edition)," which affirms the significant impact of three-dimensional visualization technology in guiding the precise diagnosis and treatment of hepatobiliary stones. The "Consensus recommendations of three-dimensional visualization for diagnosis and management of liver disease" published in an international journal demonstrates that China's research level in this field is at the forefront globally. Sioh Huang Lim et al. utilized ICG intraoperative navigation technology to visualize the extrahepatic bile ducts without radiation, enabling quicker identification of bile ducts compared to cholangiography. Liu Yangsui et al. applied fluorescence imaging technology for real-time navigation of the extrahepatic bile ducts, achieving superior outcomes in terms of surgical time, intraoperative blood loss, and postoperative hospital stay compared to the traditional surgery group. In laparoscopic re-exploration of the bile duct, Tian Guangjin et al. used ICG fluorescence navigation technology as surgical assistance, with a conversion to open surgery rate of approximately 3.3% in the navigation group compared to 22.9% in the conventional surgery group, achieving higher rates of minimally invasive abdominal surgery in the navigation group. Takeshi Aoki et al. indicated in their literature the successful staining of subsegments or liver segments in 33 out of 35 cases (94.3%) using fluorescence imaging technology for liver resection navigation. Kunshan He et al. demonstrated that near-infrared (NIR) imaging method resulted in less blood loss and shorter hospital stay compared to traditional methods. ICG fluorescence imaging technology has shown promising prospects in partial liver resection surgery. In conclusion, three-dimensional visualization technology can achieve precise preoperative differentiation of vascular variations, formulate individualized surgical plans based on reconstructed three-dimensional models, and provide real-time navigation during surgery to ensure the success of the operation. Intraoperative real-time augmented reality technology navigation helps prevent intraoperative bile duct injuries, effectively reduce severe postoperative complications, and decrease residual cysts and associated complications. Therefore, the combined application of both technologies in the treatment of choledochal cysts surgery provides better medical technological support, enhances surgical safety and precision, promotes the development of minimally invasive surgery, and holds significant clinical value.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of congenital biliary dilatation confirmed; The standard of Child-Pugh classification of preoperative liver function was; class A or B; Clinical data were complete;

Exclusion Criteria:

Patients with cardiopulmonary dysfunction who cannot tolerate surgery or anesthesia; Patients with malignant transformation; Lack of clinical data.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent choledochal dilation resection surgery from January 2010 to March 2023 in zhujiang hospital were included in this study and divided into the 3D group and non-3D group.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
CCI | Postoperative review lasted until 1 year
  Comprehensive Complication Index:integrating all recorded complications weighted by severity in a single formula.
operation time | perioperative period
  minutes
intraoperative blood loss | perioperative period
  ml

SECONDARY OUTCOMES:
Postoperative complete blood count | perioperative period
  G/L
Repeat surgery rate | perioperative period
serum bilirubin levels | perioperative period
  μmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: after 2024.5.30